CLINICAL TRIAL: NCT02408367
Title: Intensity Depended Impact of a Single Exercise Bout on Cognitive Functions in Persons With Multiple Sclerosis - a Pilot Study
Brief Title: Intensity Depended Impacts on Cognitive Functions in Persons With Multiple Sclerosis - a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jens Bansi (Other)
Responsible Party: Sponsor-Investigator, Jens Bansi, Dr Jens Bansi, Klinik Valens
Organization: Klinik Valens (Other)
Other Study IDs: KValens
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: Training; Cognition; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exercise: 30 minutes of active training at 75% of the Maximum heart rate achieved in a cardiopulmonary exercise test
  Interventions: Behavioral: Exercise; Behavioral: Relaxation
- Relaxation: 30 Minutes of passive relaxation
  Interventions: Behavioral: Exercise; Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Exercise — 30 minutes endurance training at 75% of the Maximum heart rate
Behavioral: Relaxation — 30

SUMMARY:
Multiple Sclerosis (MS) is a chronic autoimmune disease where lymphocytes inflict damage to the axons and myelin sheaths of the central nervous system. Persons with multiple sclerosis (pwMS) were long advised to avoid physical activity but the benefits of exercise to improve cardiovascular and cognitive functions in pwMS have become important aspects of standardized rehabilitation programs. Recent findings show that the achieved adaptations through exercise are associated with the intensity dependent lactate increases during exercise. This dose-response relationship between the mode and the exercise intensity implicates the relevance of the exercise protocol as higher exercise intensities seem to facilitate greater benefits, also in pwMS.

This pilot study evaluates the influences of acute bout of moderate physical exercise (cycling) and relaxation on cognitive functions at three time points.

Primary outcomes are the differences (at timepoint t2) of cognitive functions assessed via the Symbol Digit Modalities Test (SDMT) and the Brief Visuospatial Memory Test Revised (BVMT-R) T1-3 of the BICAMS battery.

Results should into a randomised controlled Trial that investigates the specific influences of a three-week training intervention on Brain-derived neurotrophic factors (BDNF), Insulin Growth Factor-1 (IGF-1) and Vascular Endothelial Growth Factor (VEGF) as central neurobiological parameters of neuroplasticity, cardiorespiratory Fitness and cognitive functions.

DETAILED DESCRIPTION:
Objectives To determine responses of an acute moderate exercise bout on cognitive functions in pwMS.

Hypothesis

* Comparisons of different Training modes: exercise (overland cycling) versus relaxation
* Improvements of cognitive functionning (Memory, processing Speed) on the Symbol Digit Modalities Test (SDMT) and the Brief Visuospatial Memory Test Revised (BVMT-R) T1-3
* Correlations between the intensity-dependent lactate increases and cognitive functions

Experimental design Two-pronged, case controlled study. Randomization of 20 MS patients into a Group "Exercise" (n=10) - that perform 30 minutes cycling on an Ergometer - or "Relaxation (n=10) that perform relaxation in a comfortable and quiet environment. Both groups crossover at t2 into the respective Group. The study is set into the normal rehabilitation program and participants are given physician clearance, are informed about the study and give their written consent before the study starts.

Cognitive assessment is performed with the Symbol Digit Modalities Test (SDMT) and the Brief Visuospatial Memory Test Revised (BVMT-R) T1-3.

SDMT tests information of processing speed. The test consists of single digits paired with abstract symbols. Rows of the nine symbols are arranged pseudo-randomly. The participant must say the number that corresponds with each symbol. The SDMT can be completed within 5 min, including instructions, practice and testing. The good psychometric properties of the SDMT are well described.

BVMT-R T1-3 requires the the participant to inspect a 2 × 3 stimulus array of abstract geometric figures. There are three learning trials of 10 s. The array is removed and the patient is required to draw the array from memory, with the correct shapes in the correct position. The psychometric properties of the BVMT-R T1-3 are good. Cognitive functions are assessed at time points t1 and t2 after Exercise / Relaxation.

At baseline participants perform a progressive cardiopulmonary exercise test (CPET) on a cycle ergometer (Ergoline 800, Germany). Cardiopulmonary fitness level was monitored by direct and continuous measurements (breath by breath) of maximum oxygen consumption (VO2peak) by ergospirometer (PanGas, CPX, Germany).

The exercise protocol consisted of (a) first 3 minutes at rest (no pedalling) on the cycle ergometer; (b) 3 minutes of unloaded pedalling as a warm up; (c) testing phase until the participant reached a symptom limited maximum. Workload was continuously ramp type increased by 5-10 Watts every minute to ensure 8-12 minutes of testing; (d) the final 3 minutes were unloaded pedalling to cool down. Heart rate (Polar Electro, Kempele, Finland) and blood pressure (Riva Rocci) were monitored for the last 10 seconds every 2 minutes during the test. The 10-point BORG scale therapy short form assessed the rate of perceived exertion (RPE) at phases (c) and (d). Peak oxygen consumption (VO2peak) was defined as the highest VO2 value when the following criteria were attained: respiratory equivalent ratio (RER) > 1.10; peak heart rate (HRpeak) within 10 min-1 of age predicted maximum and rating of exertion (RPE > 8.5).

The exercise bout consists of 30 minutes physiologically defined heart rate controlled cycling at 50-60 rounds per minutes (rpm) at the lactate threshold (equal to 75% of HRpeak or 60% VO2max).

Relaxation consists of 30 minutes resting in a comfortable and quiet surrounding. Exercise and Relaxation are performed at timepoints t1 and t2.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability status scale (EDSS) score of 1.5 - 6.0

Exclusion Criteria:

* Persisted infections, acute psychotic disorders, cardiovascular and pulmonal diseases, neuropsychological disorders that serverly impact the assessment or were psychotropic medication within the last six week.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with multiple sclerosis holding an score of 1.5-6.0 on the Expanded Disability Staus Ccale (EDSS)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Brief International Cognitive Assessment of Multiple Sclerosis (BICAMS) | 3 months
  Cognitive assessment battery consisting of Symbol Digit modality test (SDMT) and the Brief Visuospatial Memory Test Revised (BVMT-R) T1-3.

SECONDARY OUTCOMES:
Cardiorespiratory parameters | 3 months
  Resting and maximum heart rate achieved in cardiopulmonary exercise test
Lactate | 3 months
  Lactate concentrations under rest, at the thresholds (lactate and respiratory compensation Point)

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Kesselring, Univ.Prof, Principal Investigator — Kliniken-Valens, Rehabilitation-Clinic Valens
Locations (1):
- Kliniken-Valens, Valens, Canton of St. Gallen, Switzerland